# Injection Therapy in Patients with Lateral Epicondylitis

ID: 2018/12

**Document Date: 05/13/2018** 

#### INFORMED CONSENT FORM

#### Dear participant

We examine the Comparison of the Effect of Hyaluronic Acid and Prolotherapy Injection on Pain, Upper Extremity Functions and Grip Strength in Patients with Lateral Epicondylitis. The name of the study is "Comparison of the Effectiveness of Hyaluronic Acid and Prolotherapy Injections in Patients with Lateral Epicondylitis".

We suggest you to participate in this research. You are free to take part in this research or not. Participation in the study is voluntary. We would like to inform you about the research before your decision. If you want to participate in the research after reading and understanding this information, sign the form.

The reason we want to do this research is to compare the effect of hyaluronic acid and prolotherapy injection on pain, upper limb functions and grip strength. Your participation in this study, which will be held at the Inonu University Turgut Ozal Medical Center Physical Medicine and Rehabilitation Service, is important for the success of the research.

If you agree to participate in the research, Prof. Dr. You will be evaluated under the responsibility of Zühal Altay. If you are deemed appropriate after some evaluations, you will be included in this study.

Possible risks during the evaluations: Assessments to be made within the scope of the study do not contain any risks. Nevertheless, the problems and risks that may arise during the continuation of the study will be communicated to you.

You can refuse to participate in this study. You also have the right to withdraw your consent at any stage of the study (with the condition of notifying researchers in advance, without prior notice).

You will not be charged any fee to participate in this study. You will not receive an additional payment because you have participated in the study.

Medical information about you will be kept confidential, but may be reviewed, if required, by officials, ethics committees or government authorities overseeing the quality of the study.

### Statement of the Participant (Patient's Statement);

Dear Professor Dr. Zühal Altay; The above information about this research was conveyed to me by stating that a research will be conducted at the Inonu University Turgut Ozal Medical Center Physical Medicine and Rehabilitation Service. In line with this information, I was invited to the research as a "participant".

I believe that if I participate in this research, the confidentiality of my information that I should stay with the doctor will be approached with great care and respect during this research. I was given sufficient confidence that my personal information will be protected with utmost care during the use of research results for educational and scientific purposes.

I can withdraw from the research without showing any reason during the execution of the project. (However, I am aware that it would be appropriate for me to notify the advance that I will withdraw from the research in order not to leave the researchers in a difficult situation.) I can also be excluded from the research by the researcher, provided that my medical condition is not harmed.

I do not assume any monetary responsibility for the expenditures for the research. I will not receive a payment.

Necessary assurance was provided that any medical intervention would be provided if any health problems that may arise due to the research application, whether direct or indirect, occur. (I will not be under a monetary burden regarding these medical interventions.)

When I encounter a health problem during the research; at any hour, Prof. Dr. I know that I can call Zühal ALTAY on the mobile phone number 05322978238 or from the Inonu University Turgut Ozal Medical Center Physical Medicine and Rehabilitation Department.

I do not have to participate in this research and may not participate. I have not encountered compelling behavior in participating in the research.

I understand all the explanations made to me in detail. I decided to take part as a participant in this research project mentioned after a certain period of thinking on my own. I accept the invitation on this matter with great satisfaction and volunteerism.

A copy of this signed form sheet will be given to me.

| Participant; |
|--------------------|
| Name and surname: |
| Address: |
| Phone. |
| Signature: |
| Interview witness; |
| Name and surname: |
| Address: |
| Phone. |
| Phone. Signature: |

## Researcher:

Name surname, title: Dr. Hakan APAYDIN

Address: İnönü University Faculty of Medicine, Department of Physical Medicine and

Rehabilitation Tel: 05423498009

Signature: